CLINICAL TRIAL: NCT03372512
Title: Fluid Status Assessed by Bioelectrical Impedance Spectroscopy and Its Association With T1-mapping by Cardiovascular Magnetic Resonance Imaging
Brief Title: Fluid Status and T1-mapping by CMR
Acronym: BCM-CMR-T1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Andreas Kammerlander, MD, Medical University of Vienna
Other Study IDs: BCM-CMR-T1
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Heart Diseases; Heart Failure; Valvular Heart Disease
MeSH Terms: conditions — Heart Diseases; Heart Failure; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fluid overload (Liters) ≥ median
  Interventions: Diagnostic Test: Bioimpedance spectroscopy
- Fluid overload (Liters) < median
  Interventions: Diagnostic Test: Bioimpedance spectroscopy

INTERVENTIONS:
Diagnostic Test: Bioimpedance spectroscopy — Fluid overload will be assessed by bioimpedance spectroscopy
  Other Names: BCM measurement

SUMMARY:
It is unclear to what extent systemic fluid overload has an impact on T1-mapping results by cardiovascular mangetic resonance imaging.

In this study, patients will undergo body composition monitoring assessing systemic fluid overload and T1-mapping using MOLLI by cardiovacular magnetic resonance imaging in order to investigate a possible association with each other.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* patient undergoing cardiovascular magnetic resonance imaging

Exclusion Criteria:

* Unwillingness to participate
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiovascular magnetic resonance imaging including T1-mapping are invited to participate in the study where fluid status will be assessed by bioimpedance spectroscopy right before cardiovascular magnetic resonance imaging.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Native T1-mapping | baseline
  Association of fluid overload and native T1 values of left ventricular myocardium
Extracellular Volume by Cardiovascular magnetic resonance imaging | baseline
  Association of fluid overload and extracellular volume of left ventricular myocardium

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria